CLINICAL TRIAL: NCT05557097
Title: Failed Instrumental Delivery Following Combined Clinical and Intrapartum Sonographic Assessment of the Fetal Head Position vs Conventional Labor Management: Propensity Score Matched Analysis of Prospective Data From an International Dataset
Brief Title: PROPENSITY-ID: Sonographic and Clinical Assessment of Head Position Prior to Instrumental Delivery and Labour Outcomes
Acronym: PROPENSITYID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Parma (Other)
Collaborators: Monash Medical Centre (Other); University Hospital of Torrejon (Other)
Responsible Party: Sponsor
Other Study IDs: 337/2022/OSS/UNIPR
Record Dates: First submitted 2022-09-19; First posted 2022-09-27 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-06

CONDITIONS: Instrumental Delivery; NEC, Affecting Fetus or Newborn; Second Stage Cesarean Delivery; Occiput Position
Keywords: Vacuum extractor; Forceps; Vaginal examination; Intrapartum ultrasound
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group ultrasound + vaginal examination: Patients submitted to instrumental delivery by clinicians who routinely perform intrapartum sonography as an adjunct to clinical examination prior to vacuum delivery
  Interventions: Diagnostic Test: Intrapartum sonography
- Group vaginal examination: Patients submitted to instrumental delivery by clinicians not performing intrapartum sonography prior to vacuum delivery

INTERVENTIONS:
Diagnostic Test: Intrapartum sonography — Intrapartum ultrasound performed as an adjunct to clinical examination to assess fetal occiput position prior to performing vacuum delivery
  Groups: Group ultrasound + vaginal examination

SUMMARY:
Instrumental delivery is performed in 3-15% of all births (1). Successful instrumental delivery avoids need for cesarean section with associated maternal surgical morbidity, risk from neonatal disimpaction and future pregnancy implications. However, instrumental birth carries risk of maternal perineal and anal sphincter injury, postpartum haemorrhage, shoulder dystocia and fetal trauma (2,3). Additionally, failure of instrumental birth requires delivery by cesarean section with a more deeply impacted fetal head, resulting in compounding of fetal and maternal risks (3,4). Therefore, appropriately identifying women that are at risk of failed instrumental birth is important to reduce maternal and neonatal morbidity.

Fetal head position and station are key determinants in success of instrumental birth, traditionally assessed with digital vaginal examination (1,5). There is now high quality evidence showing that intrapartum ultrasound is a more reliable tool in determining fetal head position and station compared to digital vaginal examination (6,7). Additionally, intrapartum ultrasound has been shown to predict outcome of instrumental birth and improve accuracy of instrument placement (8-11).

However, no randomised studies to date have demonstrated a benefit in maternal and neonatal morbidity from using intrapartum ultrasound, possibly due to being underpowered. Low recruitment of studies has been suggested to occur due to practitioners electing to use ultrasound rather than randomise participants, despite the absence of evidence supporting clinical benefit (13).

This study aims to evaluate whether the assessment of the fetal occiput position by intrapartum sonography before instrumental delivery improves labour outcomes by using an observational design with propensity score matching analysis.

This international multicentre prospective observational study will compare outcomes of two parallel groups:

* Group 1: patients submitted to instrumental delivery preceded by the use of ultrasound for the assessment of the occiput position by clinicians who routinely perform intrapartum sonography as an adjunct to clinical examination prior to vacuum delivery
* Group 2: patients having submitted to instrumental delivery without the adjunct of by clinicians not performing intrapartum sonography prior to vacuum delivery

The investigators will perform a propensity score (PS) matching analysis to assess the effect of US as an adjunct to clinical examination prior to instrumental delivery on the occurrence of failed instrumental delivery, adjusting for important differences in baseline characteristics between groups to reduce confounding bias. The investigators will assess two primary outcomes of vaginal delivery and composite adverse perinatal outcome in additional to maternal morbidity and instrumental failure rates.

DETAILED DESCRIPTION:
Introduction Instrumental delivery is commonly performed during the second stage of labor with the aim to expedite delivery in conditions of second stage dystocia or non-reassuring fetal condition and is estimated to account for approximately 3-15% of all births. The appropriate use of vacuum extractor and forceps is crucial to avoid unnecessary and potentially challenging second-stage caesarean sections, however a 4-6% failure rate has been reported following attempted instrumental delivery. When this occurs, caesarean section is required to deliver the fetus. However, caesarean section following failed instrumental delivery is acknowledged to be associated with an increased incidence of maternal and fetal complications including neonatal trauma, skull fracture, intracranial haemorrhage, neonatal acidaemia and transfer to NICU as well as postpartum haemorrhage, surgical injury and third- or fourth-degree perineal tears compared to a successful vacuum delivery.

The decision to expedite delivery by means of caesarean section during the second stage of labor has also been associated with maternal complications including uterine incision extension, incidental cystotomy and with an increased frequency of fetal injury. Therefore, the decision as to which intervention to perform is crucial to optimize the maternal and neonatal outcomes when an obstetric intervention is indicated during the second stage of labor.

Fetal head position and station are among the major determinants of successful instrumental delivery. Instrumental delivery is recommended following the ascertainment of the fetal head position when the station is below the level of the maternal ischial spines (level 0). A secondary analysis of a randomized controlled trial conducted on a group of women submitted to instrumental vaginal delivery has shown that the risk of failed vacuum extraction is increased in the event of inaccurate placement of the instrument, which is favoured by a high fetal station and a non-occiput anterior position - i.e. a malposition - of the fetal head. Fetal head position and station have been traditionally assessed by digital examination. However, such evaluation has been shown to yield limited accuracy and poor reproducibility. Akmal et al. compared the accuracy of vaginal examination versus transabdominal sonography in the ascertainment of the head position prior to instrumental delivery showing an overall 27% rate of misdiagnosis at vaginal examination, which was mainly accounted by cases in occiput posterior position and station at the level of the ischial spines. Wong et al conduced a randomized controlled trial (RCT) on 50 patients undergoing instrumental delivery by means of vacuum extractor due to second stage dystocia by measuring distance between the centre of the cignon and the flexion point between the cases submitted (n=25) and those not submitted (n=25) to intrapartum US in addition to the vaginal examination. The mean distance was lower in the patients submitted to intrapartum sonography in addition to clinical examination compared to those who had only vaginal examination (2.1+1.3 vs 2.8+1.0 cm, p<0.05).

Conversely, intrapartum sonography has been demonstrated to be a reliable tool for the assessment of the fetal head station and position, particularly in the second stage of labor. The transabdominal approach is considered the gold standard method for the diagnosis of the occiput position, while the transperineal approach is commonly used for the objective measurement of the fetal station. The US parameters have also been shown to be more accurate than clinical examination in predicting the outcome of instrumental vaginal delivery. On this basis, the International Guidelines endorse the use of intrapartum sonography in conditions of abnormal progression of the first or of the second stage of labor and in the event of uncertainty of the occiput position following vaginal examination prior to perform an instrumental delivery.

Hypothesis and Justification for the study

While grade "A" evidence supports the role of intrapartum sonography in the ascertainment of the occiput position, to date three randomized studies as well as two systematic reviews have failed to demonstrate a role of intrapartum sonography in improving labor outcomes. This can be explained by the fact that, given the low frequency of such adverse outcomes, a large number of randomized cases is warranted to demonstrate a potential benefit of ultrasound in adjunct to clinical examination when compared to clinical examination only. Two of these studies were indeed underpowered to demonstrate clinical benefits in terms of failed instrumental delivery and perinatal outcomes. The R.I.S.POS.T.A. trial was adequately powered to investigate whether the use of intrapartum US is associated with a reduction of the frequency of failed vacuum delivery compared to standard clinical management of labor, however the study was preliminary concluded upon advice of a data safety monitoring committee based on exceedingly slow recruitment rate and an unexpectedly low frequency of failed vacuum delivery. On this basis, the Authors hypothesized that most practitioners commonly perform sonography before attempted vacuum extraction even in the absence of any evidence supporting its clinical benefit, and that randomization was considered only when the fetal extraction was considered easy.

Propensity score matching analysis allows to design and analyse an observational - i.e. non-randomized - dataset to make it mimic some of the particular characteristics of a RCT. Based on the assumption that a properly conducted RCT is highly unlikely to be feasible, the investigators hypothesize that propensity score matching analysis may allow to perform an adequately powered evaluation of the potential clinical benefits - in terms of successful instrumental delivery and maternal and fetal outcomes - of intrapartum sonography in adjunct to clinical examination compared to conventional labor management.

Study objectives

To evaluate whether the assessment of the fetal occiput position by intrapartum sonography before instrumental delivery improves labor outcome.

The two primary outcomes will be vaginal delivery and composite adverse perinatal outcome. Composite adverse perinatal outcome will be defined based on the occurrence of either shoulder dystocia, acidaemia (as defined by arterial cord pH <7.0 and/or a base excess >12.0), Apgar score <7 at 5 minutes, neonatal injury (e.g. intracranial haemorrhage, skull fracture), NICU admission, ischemic-hypoxic encephalopathy and death.

Secondary outcomes will include maternal complications including third and four-degree tear, postpartum haemorrhage and surgical injury, as well as sequential instrumental delivery by forceps.

Study design

International multicentre prospective data collection which will involve tertiary maternity units with reported instrumental delivery rates around 5% or above. A minimum number of 130 patients is expected to be collected by each participating Unit.

The study will consist in a multicentre prospective data collection of two parallel groups:

* Group 1: patients submitted to instrumental delivery preceded by the use of ultrasound for the assessment of the occiput position by clinicians who routinely perform intrapartum sonography as an adjunct to clinical examination prior to vacuum delivery
* Group 2: patients having submitted to instrumental delivery without the adjunct of by clinicians not performing intrapartum sonography prior to vacuum delivery

Patients will be counselled regarding the aim of the study on admission to the labor ward. The acquisition of verbal consent for the pseudoanonymized data collection in the event of instrumental delivery will be a prerequisite for study enrolment. Data will be prospectively collected from case notes of women submitted to instrumental delivery and sent to the coordinating centre (University of Parma) for analysis at the end of the study period.

Statistical methods

In order to reduce the impact of the important differences in baseline characteristics between the intrapartum sonography + clinical examination and the clinical examination only groups, the investigators will perform a propensity score (PS) matching analysis to assess the effect of US as an adjunct to clinical examination prior to instrumental delivery on the occurrence of failed instrumental delivery, adjusting for the confounding bias caused by this imbalance. Compared with classic multivariate adjustments, the PS permits finer adjustments for wider sets of covariates. PS will be defined as the conditional probability of having US given the measured covariates in order to balance covariates in the two groups.

To obtain the PS, a logistic regression model will be fitted with intrapartum sonography + clinical examination as the dependent variable, then the investigators will model the conditional probability of having a failed instrumental delivery as a function of baseline and those clinical characteristics associated with having a vacuum delivery. The investigators will use the PS to match, without replacement, each case of intrapartum sonography + clinical examination prior to vacuum delivery with the clinical examination only that had the closest PS in 1:1 ratio, in order to optimize the precision of the estimate of association and limit bias. The investigators will also accept cases only if the difference in PS between matched cases is small (preset caliper), to obtain a better balance between the intrapartum sonography + clinical examination group and clinical examination only group as matched samples. The investigators will compute standardized differences for all variables included in the PS before and after matching, to assess the effect of matching on the imbalance, and will aim a 10% standardized difference to be the limit for a correct balance. After matching, the investigators will compare the failed vacuum delivery rate between the intrapartum sonography + clinical examination group and the clinical examination only as matched group. Finally, the investigators will calculate the odds ratio to quantify the association between intrapartum sonography and failed vacuum delivery using univariate logistic regression analysis fitted by generalized estimating equations to account for matched data.

Sample size and power

Based on available data, the estimated failure rate of instrumental delivery ranges between 4-6%. The baseline risk of failed instrumental delivery in the control group (clinical examination only) will be estimated at around 4%. Based on the assumption that the ultrasound assessment of the fetal head position could halve the frequency of failed instrumental delivery up to 2%, the total sample size of "matched" patients required in order to obtain statistical power of 80% (P <0.05) would be 2282, i.e. 1141 cases per arm. The prospective multicentre design of the study is expected to allow the enrolment of an over two-fold higher number of cases compared to the required sample size.

Based on published data, the investigators estimate that this sample size is enough also to investigate the second primary outcome of the study, i.e. composite adverse perinatal outcome as above defined.

ELIGIBILITY:
Inclusion Criteria:

* Non-anomalous singleton pregnancies
* Cephalic presenting fetus
* Gestational age > 36+0 weeks
* Clinical indication for instrumental delivery

Exclusion Criteria:

* Any contraindication to instrumental delivery
* Maternal age <18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an international multicentre study involving tertiary maternity units with a reported instrumental delivery rate at or above 5%. Women >18 years old, with singleton pregnancies, fetus in cephalic presentation, and gestation >36 weeks admitted to labour ward will be consented for pseudoanonymized data collection in the event of instrumental delivery. Participants that proceed to have an indication for instrumental delivery will be included in the data collection
Sampling Method: Probability Sample
Enrollment: 2282 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Vaginal delivery | At time of successful birth of the neonate
  Achieve delivery of the neonate vaginally via vacuum or forceps delivery
Composite adverse perinatal outcome | up to 100 weeks after delivery
  Occurrence of either shoulder dystocia, acidaemia (as defined by cord umbilical pH <7.0 and/or a base excess >12.0), Apgar score <7 at 5 minutes, neonatal injury (intracranial haemorrhage, skull fracture), NICU admission, hypoxic-ischemic encephalopathy and death

SECONDARY OUTCOMES:
Maternal morbidity | up to 100 weeks after delivery
  Including third and four-degree tear, postpartum haemorrhage, surgical injury
Sequential instrumental delivery by forceps | up to 100 weeks after delivery
  Failed attempted delivery by vacuum extraction requiring vaginal delivery by forceps

CONTACTS AND LOCATIONS:
Locations (1):
- University of Parma, Parma, Italy

REFERENCES:
- [Background] Murphy DJ, Strachan BK, Bahl R; Royal College of Obstetricians and Gynaecologists. Assisted Vaginal Birth: Green-top Guideline No. 26. BJOG. 2020 Aug;127(9):e70-e112. doi: 10.1111/1471-0528.16092. Epub 2020 Apr 28. No abstract available. PMID 32346983
- [Background] Groutz A, Hasson J, Wengier A, Gold R, Skornick-Rapaport A, Lessing JB, Gordon D. Third- and fourth-degree perineal tears: prevalence and risk factors in the third millennium. Am J Obstet Gynecol. 2011 Apr;204(4):347.e1-4. doi: 10.1016/j.ajog.2010.11.019. Epub 2010 Dec 22. PMID 21183150
- [Background] Towner D, Castro MA, Eby-Wilkens E, Gilbert WM. Effect of mode of delivery in nulliparous women on neonatal intracranial injury. N Engl J Med. 1999 Dec 2;341(23):1709-14. doi: 10.1056/NEJM199912023412301. PMID 10580069
- [Background] Le Brun C, Beucher G, Morello R, Jones F, Lamendour N, Dreyfus M. [Failure of vacuum extractions: risk factors, maternal and fetal issues]. J Gynecol Obstet Biol Reprod (Paris). 2013 Nov;42(7):693-702. doi: 10.1016/j.jgyn.2013.04.003. Epub 2013 May 20. French. PMID 23702434
- [Background] Ramphul M, Kennelly MM, Burke G, Murphy DJ. Risk factors and morbidity associated with suboptimal instrument placement at instrumental delivery: observational study nested within the Instrumental Delivery & Ultrasound randomised controlled trial ISRCTN 72230496. BJOG. 2015 Mar;122(4):558-63. doi: 10.1111/1471-0528.13186. Epub 2014 Nov 21. PMID 25414081
- [Background] Dupuis O, Silveira R, Zentner A, Dittmar A, Gaucherand P, Cucherat M, Redarce T, Rudigoz RC. Birth simulator: reliability of transvaginal assessment of fetal head station as defined by the American College of Obstetricians and Gynecologists classification. Am J Obstet Gynecol. 2005 Mar;192(3):868-74. doi: 10.1016/j.ajog.2004.09.028. PMID 15746684
- [Background] Akmal S, Kametas N, Tsoi E, Hargreaves C, Nicolaides KH. Comparison of transvaginal digital examination with intrapartum sonography to determine fetal head position before instrumental delivery. Ultrasound Obstet Gynecol. 2003 May;21(5):437-40. doi: 10.1002/uog.103. PMID 12768552
- [Background] Wong GY, Mok YM, Wong SF. Transabdominal ultrasound assessment of the fetal head and the accuracy of vacuum cup application. Int J Gynaecol Obstet. 2007 Aug;98(2):120-3. doi: 10.1016/j.ijgo.2007.05.021. Epub 2007 Jun 22. PMID 17585916
- [Background] Ghi T, Eggebo T, Lees C, Kalache K, Rozenberg P, Youssef A, Salomon LJ, Tutschek B. ISUOG Practice Guidelines: intrapartum ultrasound. Ultrasound Obstet Gynecol. 2018 Jul;52(1):128-139. doi: 10.1002/uog.19072. PMID 29974596
- [Background] Kahrs BH, Usman S, Ghi T, Youssef A, Torkildsen EA, Lindtjorn E, Ostborg TB, Benediktsdottir S, Brooks L, Harmsen L, Romundstad PR, Salvesen KA, Lees CC, Eggebo TM. Sonographic prediction of outcome of vacuum deliveries: a multicenter, prospective cohort study. Am J Obstet Gynecol. 2017 Jul;217(1):69.e1-69.e10. doi: 10.1016/j.ajog.2017.03.009. Epub 2017 Mar 19. PMID 28327433
- [Background] Bultez T, Quibel T, Bouhanna P, Popowski T, Resche-Rigon M, Rozenberg P. Angle of fetal head progression measured using transperineal ultrasound as a predictive factor of vacuum extraction failure. Ultrasound Obstet Gynecol. 2016 Jul;48(1):86-91. doi: 10.1002/uog.14951. Epub 2016 Jun 10. PMID 26183426
- [Background] Ramphul M, Ooi PV, Burke G, Kennelly MM, Said SA, Montgomery AA, Murphy DJ. Instrumental delivery and ultrasound : a multicentre randomised controlled trial of ultrasound assessment of the fetal head position versus standard care as an approach to prevent morbidity at instrumental delivery. BJOG. 2014 Jul;121(8):1029-38. doi: 10.1111/1471-0528.12810. Epub 2014 Apr 11. PMID 24720273
- [Background] Ghi T, Dall'Asta A, Masturzo B, Tassis B, Martinelli M, Volpe N, Prefumo F, Rizzo G, Pilu G, Cariello L, Sabbioni L, Morselli-Labate AM, Todros T, Frusca T. Randomised Italian Sonography for occiput POSition Trial Ante vacuum (R.I.S.POS.T.A.). Ultrasound Obstet Gynecol. 2018 Dec;52(6):699-705. doi: 10.1002/uog.19091. Epub 2018 Nov 8. PMID 29785716
- [Background] Barros JG, Afonso M, Martins AT, Carita AI, Clode N, Ayres-de-Campos D, Graca LM. Transabdominal and transperineal ultrasound vs routine care before instrumental vaginal delivery - A randomized controlled trial. Acta Obstet Gynecol Scand. 2021 Jun;100(6):1075-1081. doi: 10.1111/aogs.14065. Epub 2021 Jan 12. PMID 33319355
- [Background] Bellussi F, Di Mascio D, Salsi G, Ghi T, Dall'Asta A, Zullo F, Pilu G, Barros JG, Ayres-de-Campos D, Berghella V. Sonographic knowledge of occiput position to decrease failed operative vaginal delivery: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2022 Apr;226(4):499-509. doi: 10.1016/j.ajog.2021.08.057. Epub 2021 Sep 4. PMID 34492220
- [Background] Mappa I, Tartaglia S, Maqina P, Makatsariya A, Ghi T, Rizzo G, D'Antonio F. Ultrasound vs routine care before instrumental vaginal delivery: A systematic review and meta-analysis. Acta Obstet Gynecol Scand. 2021 Nov;100(11):1941-1948. doi: 10.1111/aogs.14236. Epub 2021 Aug 8. PMID 34314520
- [Background] Ghi T, Youssef A. Does ultrasound determination of fetal occiput position improve labour outcome? BJOG. 2014 Sep;121(10):1312. doi: 10.1111/1471-0528.12956. No abstract available. PMID 25155321
- [Background] Dall'Asta A, Rizzo G, Ghi T. Intrapartum ultrasound before instrumental vaginal delivery: Clinical benefits are difficult to demonstrate. Acta Obstet Gynecol Scand. 2021 May;100(5):988-989. doi: 10.1111/aogs.14082. Epub 2021 Feb 5. No abstract available. PMID 33423283